CLINICAL TRIAL: NCT00798122
Title: Study of Women With Acute Coronary Syndromes and Nonobstructive Coronary Artery Disease
Acronym: SWAN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 07-050; DD CSDA 2006066 (Other Grant/Funding Number: DORIS DUKE CHRTBL FND)
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Acute Coronary Syndromes
Keywords: sex; acute coronary syndromes; normal angiogram; no obstruction at angiography; women
MeSH Terms: conditions — Acute Coronary Syndrome; Coitus | interventions — Ultrasonography, Interventional

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women (Experimental): IVUS and MRI performed in women with no obstructive CAD at angiography
  Interventions: Procedure: Intravascular ultrasound; Procedure: MRI

INTERVENTIONS:
Procedure: Intravascular ultrasound — intravascular ultrasound
Procedure: MRI — cardiac MRI

SUMMARY:
Approximately 600,000 women are treated for acute coronary syndrome (ACS) annually in the US. ACS includes heart attack and a milder form called unstable angina. Many of these women have angiograms of which 14-39% show no "significant" coronary artery disease (CAD, cholesterol plaque accumulation in arteries of the heart). The remaining majority of women with ACS have cholesterol plaque buildup which appears severe enough on angiography to limit blood flow to the heart.

It is difficult to advise women with heart attacks and no major heart artery blockages on what to do if chest pain happens again. Additional studies are needed to find out why this sort of heart attack happens and to help doctors understand how to treat patients who have this problem in the best possible way.

Some women with heart attacks who have no major blockage in heart arteries have cholesterol plaque in the arteries of the heart cannot be seen on angiography but can be seen using a newer technique called intravascular ultrasound (IVUS). IVUS involves creating pictures of the artery walls using ultrasound (sound waves) from within the artery itself. In some women without major heart artery blockage, heart attack is caused by low blood flow due to disease of smaller blood vessels which cannot be seen on angiography or IVUS. This problem can be found using magnetic resonance imaging (MRI), which can show blood flow to the heart. MRI may also be used to show where the heart has been damaged. The pattern of damage could suggest that a heart attack in a woman, who has no badly blocked heart arteries, happened for one (or more) of these reasons or another reason.

The Study of Women with ACS and Non-obstructive CAD (SWAN) will use IVUS and MRI to help determine the reasons for heart attacks in women with no major blockages in heart arteries.

ELIGIBILITY:
Inclusion Criteria:

* women
* positive cardiac markers and/or ST elevation
* scheduled for angiography

Exclusion Criteria:

* prior diagnosis of obstructive CAD
* contraindication to IVUS and/or MRI
* use of vasospastic agent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-03-01 (Actual); Primary Completion 2011-09-06 (Actual); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
IVUS and MRI findings | within one week of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Harmony Reynolds, M.D., Principal Investigator — NYU Langone Health
Locations (1):
- NYU Medical Center and Bellevue Hospital Center, New York, New York, United States

REFERENCES:
- [Derived] Reynolds HR, Srichai MB, Iqbal SN, Slater JN, Mancini GB, Feit F, Pena-Sing I, Axel L, Attubato MJ, Yatskar L, Kalhorn RT, Wood DA, Lobach IV, Hochman JS. Mechanisms of myocardial infarction in women without angiographically obstructive coronary artery disease. Circulation. 2011 Sep 27;124(13):1414-25. doi: 10.1161/CIRCULATIONAHA.111.026542. Epub 2011 Sep 6. PMID 21900087